CLINICAL TRIAL: NCT05288244
Title: The Effect of Foot Bath and Lavender Oil Sniffing on the Severity of Insomnia in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Furkan Şahin, principal investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EO-F-SAHIN-001
Record Dates: First submitted 2022-02-09; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Cancer Patient

STUDY DESIGN:
Intervention Model Description: randomization controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- foot bath (Experimental): It will be applied to the patients in group A (foot bath) every evening between 21.00-21.20 for 14 days. The steps of the procedure are as follows:
  * To be used in the footbath, a footbath tub, water at 38-40°C, a thermometer to measure the temperature of the water, foot towels, clean socks, gloves are prepared.
  * With the water temperature adjustment button in the foot bath tub, wait until the temperature of the water reaches 38-40 °C
  * Between 21:00 and 21:20, the feet are kept in water with a constant temperature of 38-40 °C for 20 minutes. (While the process is in progress, the water temperature is checked intermittently with a laser thermometer.)
  Interventions: Other: To evaluate the effect of foot bath applied for 2 weeks on insomnia in cancer patients.
- lavender oil snuff (Experimental): The L group (lavender oil sniffing) will be applied, the lavender oil sniffing process will be applied every evening between 21.00-21.05 for 14 days, and the process steps will be as follows;
  * Essential lavender oil to be used for the enterprise is obtained from a company that has business registration and TS EN ISO 9001: 2008 quality certificates with the number G06-3231 from the Ministry of Food, Agriculture and Livestock.
  * 3 drops of the obtained lavender oil are dripped onto the cotton pad.
  * The prepared cotton pad is fixed on the patient's clothing in the upper chest and shoulder area with a locked needle and the patient is asked to sniff for 5 minutes (Özkaraman et al., 2018).
  Interventions: Other: To evaluate the effectiveness of smelling lavender oil applied to cancer patients for 2 weeks on sleep.
- foot bath and lavender oil snuff (Experimental): AL group (both foot bath and lavender oil sniffing),for 14 days, every evening between 21.00-21.20, foot bath and lavender oil sniffing between 21.00-21.05 will be applied together.
  Interventions: Other: To evaluate the effect of foot bath and lavender oil applied for 2 weeks on insomnia in cancer patients.

INTERVENTIONS:
Other: To evaluate the effect of foot bath applied for 2 weeks on insomnia in cancer patients. — To evaluate the effect of foot bath applied for 2 weeks on insomnia in cancer patients.
  Arms: foot bath
Other: To evaluate the effectiveness of smelling lavender oil applied to cancer patients for 2 weeks on sleep. — To evaluate the effectiveness of smelling lavender oil applied to cancer patients for 2 weeks on sleep.
  Arms: lavender oil snuff
Other: To evaluate the effect of foot bath and lavender oil applied for 2 weeks on insomnia in cancer patients. — To evaluate the effect of foot bath and lavender oil applied for 2 weeks on insomnia in cancer patients.
  Arms: foot bath and lavender oil snuff

SUMMARY:
Insomnia is observed due to the cancer itself, the treatments applied and the complaints experienced. Insomnia disrupts comfort and reduces the quality of life. This work; It is planned to evaluate the effect of foot bath and lavender oil scent applied for 14 days on the severity of insomnia.

Within the scope of the study, the participants will be divided into three groups and the procedures will be applied. In the first group, between 21:00 - 21:20, you will be asked to place your feet in the foot bath apparatus with 38-40 ° C warm water. In the second group, between 21:00 and 21:05, a cotton pad with three drops of pure lavender oil will be fixed on the clothes in the upper chest and shoulder area, and you will be able to smell it for 5 minutes. The third group will be given both a foot bath and a scent of lavender oil.Which group the patients will fall into will be determined randomly.

Research hypotheses:

H0-1: Foot bath has no effect on the severity of insomnia in cancer patients. H1-1: Foot bath has an effect on the severity of insomnia in cancer patients H0-2: Smelling lavender oil has no effect on the severity of insomnia in cancer patients.

H1-2: Smelling lavender oil has an effect on the severity of insomnia in cancer patients.

H2: The effect of foot bath and lavender oil scenting applied together on the severity of insomnia in cancer patients is more than the application of only foot bath.

H3: Foot bath and lavender oil sniffing applied together has a greater effect on the severity of insomnia in cancer patients than only lavender oil sniffing.

DETAILED DESCRIPTION:
Cancer, which is increasing day by day in the world, is the most common cause of death after cardiovascular diseases. One out of every six deaths in the world and one in five deaths in our country is caused by cancer. Cancer itself and its treatment cause physical, psycho-social problems that negatively affect the quality of life of individuals during the disease process. Among these symptoms are cognitive and psychological disorders, especially pain, fatigue, sleep problems, loss of appetite, weight loss, shortness of breath, skin changes, weakness, nausea-vomiting, etc.Fatigue and insomnia, which are common in cancer patients, can be seen as a result of pain and fatigue, and chemotherapy and radiotherapy applied to patients also trigger this situation.Sleep problems are a condition that causes discomfort in the quality and quantity of the resting order and affects the lifestyle and quality of the individual.Although it is a common problem in cancer patients, it is among the neglected symptoms. The causes of sleep problems include the type and stage of the disease, the drug treatments used, accompanying emotional problems such as fatigue, pain, vomiting, shortness of breath, loss of appetite, constipation, and depressive mood and not reporting sleep problems in cancer patients with the belief that it is commonplace.Insomnia, which is the most common sleep problem, is usually associated with some symptoms rather than being a stand-alone symptom in cancer patients. In a study, it was reported that 50% of cancer patients had sleep disorders and this situation was more common in women than men.In another study detected sleep problems in 2/3 of cancer patients and concluded that 69.4% of them had low sleep quality. In another study, on the other hand, stated that 34.4% of lung cancer patients have sleep problems at night.In another study, 36.7% of patients who received chemotherapy before treatment; 13.3% of sleep problems were detected after the sixth cure.For this reason, sleep problems in cancer patients should be questioned and managed.Cognitive-behavioral therapy, stimulus control, relaxation techniques, yoga, tai-chi, reiki, listening to music, bright white light application in the nursing management of sleep problems of cancer patients. There are applications such as aromatherapy and foot baths.Foot bath; It is a non-drug method in which different applications such as water or steam are used by nurses to protect the health of patients and help them relax. In this method, relaxation is provided and the patient's sleep quality is increased by keeping the feet at a temperature between 40-43°C for about 10-30 minutes.In another study stated that footbath at 41-42 °C applied to patients receiving chemotherapy reduces the level of fatigue and improves sleep quality. In another study, footbath with water at 38-42 °C reduced the pain of patients and allowed them to relax.Foot bath has many positive physiological effects. It is known that a water temperature of 38-40°C causes vasodilation with a parasympathetic effect, decreases vascular resistance, increases blood flow to the tips of the toes and creates relaxation in the muscles.

Florance Nightingale emphasized the importance of a healthy environment for patients and recommended the use of fragrant flowers with a high aromatherapy effect in creating this environment.Aromatherapy is the use of aromatic oils obtained from plant extracts for psychological or physical therapy.The components in these oils act by being absorbed by touch, vaginal or anal suppositories, mouth and inhalation. Aromatherapy applied through inhalation affects the individual positively in many ways, including spiritual, physical and psychological. Lavender used for this purpose is used for therapeutic purposes to provide spiritual comfort, physical and emotional well-being, and to regulate sleep disorders.In another study, it was determined that the trait anxiety of cancer patients who smelled lavender for 5 minutes before going to bed decreased and their sleep quality increased.In another study reported that aromatherapy massage reduces pain and improves the sleep quality of patients.In another study stated that inhalation of lavender oil reduces heart rate, respiratory rate and body temperature, and provides relaxation.In another study examined the effect of inhaled lavender scent on sleep in hemodialysis patients; The patients left lavender oil 15-20 cm away from the pillow by dripping two drops on the cotton in the box 30 minutes before going to sleep for a week. At the end of one week, an increase in the sleep quality of the patients was observed.

The population of the research will consist of patients hospitalized in Eskişehir City Hospital Palliative Service and Medical Oncology Service due to cancer diagnosis. The sample is the patients who meet the sample selection criteria in the specified population.

Sample selection criteria;

* over 18 years old
* Diagnosed with cancer,
* Having a sense of smell,
* Foot skin integrity is complete,
* Conscious,
* Patients who agreed to participate in the study Exclusion criteria from the study;
* Peripheral vascular disease,
* Having asthma,
* Known allergy history,
* Using products such as antiperspirants, perfumes, sprays that contain any odor on their hair and body before the procedure,
* Cancer patients receiving drug therapy for insomnia will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* Diagnosed with cancer,
* Having a sense of smell,
* Foot skin integrity is complete,
* Conscious,
* Patients who agreed to participate in the study

Exclusion Criteria:

* with peripheral vascular disease,
* with asthma,
* Known allergy history
* Before the procedure, using products such as antiperspirants, perfumes, sprays that contain any odor on their hair and body,
* Cancer patients receiving drug therapy for insomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The effect of foot bath and lavender oil scent on insomnia severity in cancer patients | first day
  Insomnia severity index and MD Anderson Symptom Index will be used to determine the severity of insomnia of the patients.
  Insomnia Severity Index consists of 7 questions. Scoring ranges from 0 to 28. While 28 points is the upper limit, it indicates that the patient has severe insomnia, while a lower score of 0 indicates that the patient does not have insomnia. The MD Anderson Symptom Index, on the other hand, is a scale used to evaluate the symptoms of the patient, consisting of a total of 19 questions. Although each question parameter is scored between 0 and 10, a score of 0 indicates that the patient has no symptoms, while the upper limit of 10 points indicates that the patient has severe symptoms.

SECONDARY OUTCOMES:
The effect of foot bath and lavender oil scent on insomnia severity in cancer patients | fiveteen day
  Insomnia severity index and MD Anderson Symptom Index will be used to determine the severity of insomnia of the patients.
  Insomnia Severity Index consists of 7 questions. Scoring ranges from 0 to 28. While 28 points is the upper limit, it indicates that the patient has severe insomnia, while a lower score of 0 indicates that the patient does not have insomnia. The MD Anderson Symptom Index, on the other hand, is a scale used to evaluate the symptoms of the patient, consisting of a total of 19 questions. Although each question parameter is scored between 0 and 10, a score of 0 indicates that the patient has no symptoms, while the upper limit of 10 points indicates that the patient has severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir City Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] -Lee, K., Cho, M., Miaskowski, C., Dodd, M. Impaired sleep and rhythms in persons with cancer. Sleep Med Rev;2004;8(3):199-212. CrossRef -Hagar, F.S. Effect of warm water foot bath on fatigue in patients undergoing hemodialysis. International Journal of Nursing Didactics,2018; 8, 26-32. -Yang, H.-L., et al. The effects of warm-water footbath on relieving fatigue and insomnia of the gynecologic cancer patients on chemotherapy. Cancer nursing,2010; 33(6): 454-460. -Yamamoto, K., Nagata,S. Physiological and psychological evaluation of the wrapped warm footbath as a complementary nursing therapy to induce relaxation in hospitalized patients with incurable cancer: a pilot study. Cancer nursing, 2011;34(3): 185-192. -Harada, T., Iwakawa, Y., Ikeda, H.Thermographic study on the preservability of heat effects of footbath with salt. Hiroshima J Med Sci, 2014;63(1-3): 1-5. -Seyyedrasooli, A., Valizadeh, L., Zamanzadeh, V., Nasiri, K., Kalantri, H. The effect of footbath on sleep quality of the elderly: A blinded randomized clinical trial. Journal of Caring Sciences, 2013; 2(4): 305-311 -Bensouilah, J. The history and development of modern-British aromatherapy. International Journal of Aromatherapy,2005; 15(3), 134-140. -Keville, K., Green, M. (2009). Aromatherapy: A Complete Guide to the Healing Art (2nd ed.). New York: Crossing Press.